CLINICAL TRIAL: NCT02670148
Title: Assessment of Chiropractic Treatment: Strength and Balance
Acronym: ACT3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ian Coulter (Other)
Collaborators: Palmer College of Chiropractic (Other); Samueli Institute for Information Biology (Other)
Responsible Party: Sponsor-Investigator, Ian Coulter, Principal Investigator, RAND
Organization: RAND (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0159
Record Dates: First submitted 2015-12-15; First posted 2016-02-01 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2018-12

CONDITIONS: Low Back Pain
Keywords: Chiropractic Manipulative Therapy; Low back pain; Trunk muscle strength; Balance; Active military personnel
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chiropractic Care (CC) (Experimental): Participants in the CC group will receive evaluation and treatment (chiropractic manipulative therapy) from a doctor of chiropractic over a 4 week period.
  Interventions: Procedure: Chiropractic manipulative therapy
- Waitlist control group (WC) (No Intervention): Participants allocated to the waitlist control group will not receive any chiropractic treatment during the active study period. These individuals will be scheduled for one additional study visit following allocation. This final study visit will be scheduled 4 weeks after allocation (± 7 days). WC participants are not restricted from receiving any other healthcare during study participation. However, participants in the WC group will be asked not to receive any chiropractic care or spinal manipulation by any other provider during the 4 week intervention period. After WC participants complete the final study visit, they will be offered chiropractic care. This treatment will not be part of the study and no data will be collected at these visits.

INTERVENTIONS:
Procedure: Chiropractic manipulative therapy — We will set an a priori treatment schedule of 8 visits at a frequency of 2 visits per week over a 4 week period. CC participants will receive chiropractic manipulative therapy (CMT). CMT procedures can be broadly divided into two types, thrust and non-thrust. Thrust CMT is a high-velocity low-amplitude procedure characterized by a single, short duration thrust (ranging from 100 to 500 ms) of low amplitude force applied to a target joint that often results in an audible sound, or cavitation. Non-thrust CMT employs low-velocity and often repeated joint movements of varying amplitude. In the event that no CMT treatment is clinically indicated, treatment will not be provided.
  Other Names: Spinal manipulative therapy
  Arms: Chiropractic Care (CC)

SUMMARY:
This study is a randomized controlled trial designed to compare the effects of 4 weeks of chiropractic care to a waitlist control group on measures of strength, balance, and endurance in military personnel experiencing non-surgical low back pain.

DETAILED DESCRIPTION:
This study will assess three functional outcomes (strength, balance and endurance) and patient-reported outcomes in participants with low back pain (LBP) treated with chiropractic care, providing evidence that may enhance our understanding of the relationship between functional outcomes and chiropractic care. The findings from this study may support the use of chiropractic care for military personnel as an effective, conservative treatment for low back pain that may also help preserve or improve functional outcomes and thus, allow active duty personnel to better perform the physical demands required of them.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18 - ≤ 40, inclusive
2. Able to provide written informed consent
3. Self-reported acute, subacute or chronic LBP at initial screen and baseline visit 1. Pain intensity of ≥ 2 on NRS within the past 24 hours.
4. Active duty status

Exclusion Criteria:

1. Any chiropractic care within 30 days of informed consent
2. Any LBP confirmed or suspected to arise from a visceral source
3. Spinal pathology or any other condition(s) contraindicating SM
4. LBP for which specific treatments outside those available within study parameters are indicated
5. Any spinal fracture within the past 6 months
6. Any spinal surgery within the past 6 months
7. LBP with positive neurologic signs indicating spinal nerve root compression, or LBP with presumptive or confirmed spinal nerve root compression
8. Imaging evidence of neuroforaminal or spinal canal stenosis or the clinical presentation of neurogenic claudication
9. Chronic pain syndrome diagnosis
10. Diagnosis or suspected systemic inflammatory arthropathy of the spine
11. Referral needed to evaluate or treat an urgent or emergent condition or to determine the status of a condition that pertains to eligibility
12. Unable to safely perform strength, balance, or endurance tests, or the ability to assess health status
13. Pregnant or planning to become pregnant within the next 6 weeks
14. Knowledge of impending transfer or absence during study period
15. Seeking or referred for Medical Evaluation Board / Physical Evaluation Board disability status (to ensure safety while performing study tests and to avoid confounding due to the potential for competing recovery goals)
16. Unable or unwilling to comply with study protocols
17. Patellar height is <15 inches or >25.5 inches

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2016-04; Primary Completion 2019-02-14 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Isometric muscle strength test using force transducer | Baseline and week 4
  During the isometric muscle strength test, participants will first be placed in a safety harness and instructed into a proper lifting position. Participants will then be instructed to pull up (with gradually increasing effort levels) against a handle attached to a force transducer with a metallic chain. Participants will be instructed to immediately stop pulling on the handle if they experience any increased discomfort. The maximum pulling force recorded during the 3 tests will be used for data analysis, and these measurements will be taken at the first and last study visit. The outcome will be the change in strength following the 4-week intervention period.

SECONDARY OUTCOMES:
One-Leg Standing Test (Stork test) via computer-activated timer | Baseline and week 4
  Participants will wear a safety harness and be instructed to remove their shoes, place their hands on their hips, and position their dominant foot against their supporting leg. The participant will then be asked to balance in the described position and raise their heel off the floor. A computer-activated timer connected to a sensor pad on the floor will start as the heel is raised. The timer will stop when the heel of the supporting foot or the other foot touches the floor. The longest holding time under conditions where the participant's eyes are open and closed will be used for data analysis. Measurements will be taken at the first and last study visit, and the outcome will be the change in balance following the intervention period.
Stopwatch-timed trunk muscle endurance assessment (Biering-Sorensen test) | Baseline and week 4
  The test is performed with a participant lying prone on a padded table. The edge of the table is aligned with the top of the pelvis leaving the head, shoulders, and trunk extending over the edge, supported by the forearms resting on a padded cushion. The lower extremities are strapped to the table as firmly as comfort will allow. The participant is instructed to lift their arms off the support while maintaining a neutral trunk position and hold the posture for as long as possible. They are instructed to end the test if they experience pain or discomfort or are unable to maintain the posture. The length of time (in seconds) the participant holds the posture is recorded (using a hand-held stopwatch) as the test length. Measurements will be taken at the first and last study visit, and the outcome will be the change in endurance following the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Coulter, PhD, Principal Investigator — RAND
Locations (1):
- Naval Branch Health Clinic, NATTC, Pensacola, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vining R, Minkalis A, Long CR, Corber L, Franklin C, Gudavalli MR, Xia T, Goertz CM. Assessment of chiropractic care on strength, balance, and endurance in active-duty U.S. military personnel with low back pain: a protocol for a randomized controlled trial. Trials. 2018 Dec 5;19(1):671. doi: 10.1186/s13063-018-3041-5. PMID 30518400